CLINICAL TRIAL: NCT02550483
Title: Novel Metabolites of Beta-Carotene and Lycopene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HS51
Record Dates: First submitted 2015-09-08; First posted 2015-09-15 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Healthy
Keywords: Healthy volunteers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Beta-Carotene Tomato Juice (Active Comparator): Participants will receive high beta-carotene tomato juice daily as part of controlled diet (base diet + high beta-carotene tomato juice).
  Interventions: Other: Base diet + high beta-carotene tomato juice
- Lycopene Tomato Juice (Active Comparator): Participants will receive high lycopene tomato juice daily as part of controlled diet (base diet + high lycopene tomato juice).
  Interventions: Other: Base diet + high lycopene tomato juice
- Placebo Beverage (Placebo Comparator): Participants will receive placebo beverage daily as part of controlled diet (base diet + placebo beverage).
  Interventions: Other: Base diet + placebo beverage

INTERVENTIONS:
Other: Base diet + high beta-carotene tomato juice — Participants will receive high beta-carotene tomato juice daily in addition to the base diet. Meals will be prepared using traditional American foods with a macronutrient composition representative of a typical American diet. The base diet will be low in betacarotene and lycopene (no carrots, sweet potato, tomatoes, and dark greens). During the controlled diet period, participants will be instructed to eat all foods and only foods provided to them, with the exception of water, coffee, tea, and diet soda.
  Arms: Beta-Carotene Tomato Juice
Other: Base diet + high lycopene tomato juice — Participants will receive high lycopene tomato juice daily in addition to the base diet. Meals will be prepared using traditional American foods with a macronutrient composition representative of a typical American diet. The base diet will be low in betacarotene and lycopene (no carrots, sweet potato, tomatoes, and dark greens). During the controlled diet period, participants will be instructed to eat all foods and only foods provided to them, with the exception of water, coffee, tea, and diet soda.
  Arms: Lycopene Tomato Juice
Other: Base diet + placebo beverage — Participants will receive a placebo beverage daily in addition to the base diet. Meals will be prepared using traditional American foods with a macronutrient composition representative of a typical American diet. The base diet will be low in betacarotene and lycopene (no carrots, sweet potato, tomatoes, and dark greens). During the controlled diet period, participants will be instructed to eat all foods and only foods provided to them, with the exception of water, coffee, tea, and diet soda.
  Arms: Placebo Beverage

SUMMARY:
The study (n = 36) will be a parallel design and will be 6 weeks in duration. Participants will start with a 2-week free-living wash-in period where they will be asked to avoid certain carotenoid-rich foods, followed by 4 weeks of a completely controlled diet. In addition to the controlled diet, participants will consume one of three beverages (300 mL/day; n = 12/group): placebo beverage (control), high beta-carotene tomato juice, and high-lycopene tomato juice. Blood, urine and feces will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* Age less than 21 or greater than 75 years
* Glucose > 126 mg/dl
* Triglycerides > 300 mg/dl
* Known allergy or intolerance to tomatoes or tomato products
* Pregnant, lactating, or intend to become pregnant during the study period
* History of bariatric surgery or nutrient malabsorption disease (such as celiac disease) or other metabolic disorders requiring special diet recommendations
* Smoker or use of tobacco products
* Presently have cancer
* Use of certain medications (prescription or over-the-counter) that may interfere with the study objectives
* Type 2 diabetes
* Use of blood-thinning medications such as Coumadin (warfarin), Dicumarol, or Miradon (anisindione)
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in apocarotenoid concentrations will be measured in blood | Baseline, 2 weeks, 4 weeks
  Apocarotenoid concentrations will be measured in blood (baseline, after washout; 2 wks; 4 wks).
Change in carotenoid concentrations will be measured in blood | Baseline, 2 weeks, 4 weeks
  Carotenoid concentrations will be measured in blood (baseline, after washout; 2 wks, 4 wks).

SECONDARY OUTCOMES:
Change in global gene expression | Baseline, 4 weeks
  Amounts of messenger RNA will be measured in blood samples to determine if the consumption of carotenoid-rich foods will affect gene expression of pathways related to cancer risk.
Change in proportion of phyla of colonic microbiota | Baseline, 4 weeks
  Ribosomal RNA will be measured to determine relative amounts of different bacterial phyla present in the colon after consumption of the juice products differing in carotenoid concentration.
Identification of unknown urinary carotenoid metabolites | Baseline, 2 weeks, 4 weeks
  Identify previously unknown carotenoid metabolites in urine.

CONTACTS AND LOCATIONS:
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

REFERENCES:
- [Derived] Cooperstone JL, Novotny JA, Riedl KM, Cichon MJ, Francis DM, Curley RW Jr, Schwartz SJ, Harrison EH. Limited appearance of apocarotenoids is observed in plasma after consumption of tomato juices: a randomized human clinical trial. Am J Clin Nutr. 2018 Oct 1;108(4):784-792. doi: 10.1093/ajcn/nqy177. PMID 30239552